CLINICAL TRIAL: NCT06535516
Title: TRANSFORM: Translational Research That Adapts New Science FOR Maltreatment Prevention Project 3
Brief Title: Resilient Roots: Supporting Youth and Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sheree Toth, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2P50HD096698 (NIH); 2P50HD096698-06 (NIH)
Record Dates: First submitted 2024-07-17; First posted 2024-08-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Trauma-Focused Cognitive Behavioral Therapy and Socialization
Who Masked: Outcomes Assessor
Masking Description: Research assistants will be blind to which arm the participant has been randomly assigned to and to study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) (Active Comparator): TF-CBT will be administered as typically implemented at Pediatric Behavioral Health and Wellness outpatient clinic
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)
- Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) and Socialization (Experimental): TF-CBT will be implemented enhanced with socialization components
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT); Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) augmented with Socialization (S)

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) — TF-CBT is a well-established trauma treatment for children ages 3-17 years that demonstrates improved outcomes relative to other active treatments. Originally developed for treatment of childhood sexual abuse, evidence from numerous randomized clinical trials (RCT) demonstrates that TF-CBT is one of the most effective treatments for children with PTSD and/or depression resulting from many forms of child abuse and neglect as well as other traumatic experiences.TF-CBT is rated by California Evidence-Based Clearinghouse for Child Welfare as highly relevant for child welfare and well-supported in improving children's outcomes, including reduced PTSD symptoms, behavior problems, depression, and shame, and improving parental support related to their children's experiences.
Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) augmented with Socialization (S) — The study will compare standard TF-CBT with TF-CBT augmented with Socialization enhancements. TF-CBT+S includes enhancements to address socioecological stress and trauma and provide coping strategies to support positive socialization.
  Arms: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) and Socialization

SUMMARY:
Resilient Roots is integrated into the TRANSFORM Center to promote translation of research findings into clinical interventions, to inform the next generation of research on child abuse and neglect (CAN), and to facilitate dissemination of research and practice knowledge/skills to varied stakeholders. Exposure to CAN frequently results in long-term detrimental effects on mental health. For youth who have experienced socioecological stress, the trauma associated with CAN may be compounded by stress and trauma deriving from experiences of stress in their communities. Interventions to address specific socioecological stress for symptomatic youth receiving human centered mental health services are lacking, and use of mental health services that are acceptable to families are too often misaligned with their representation in the population in general and overrepresentation in the child welfare system specifically. Incorporating support for families in enhancing socialization and coping skills specific to addressing contextual stress and trauma has relevance for public health. Although Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) is an evidence-based treatment for children who have experienced CAN, determining best practices for implementing enhanced TF-CBT with socialization components is urgently needed to address these gaps and provide optimal intervention. Resilient Roots is a pilot study within a RE-AIM/PRISM framework (including Reach, Effectiveness, Adoption, Implementation, and Maintenance with emphasis on contextual factors at multiple levels of the implementation setting) that will incorporate stakeholder perspectives and evaluate the incorporation of socialization into enhanced TF-CBT, while identifying barriers and facilitators to implementation to guide future larger-scale trials.

DETAILED DESCRIPTION:
Child abuse and neglect (CAN) represents a pathogenic relational environment that confers significant risk for maladaptation. The deleterious sequelae accompanying child abuse and neglect result in adverse physical and mental health consequences during childhood and initiate a negative developmental cascade that continues throughout the life course. The proximal environment involving the nuclear family, as well as more distal factors associated with the community and context, transact to undermine normal biological and psychological developmental processes in these vulnerable children. For youth from high-risk communities, these negative sequelae are compounded by the effects of additional socioecological stress that may further undermine their wellbeing and adaptive functioning. Some youth are disproportionately represented within Child Protective Services (CPS) and child welfare systems and yet less likely to receive mental health services, particularly high-quality evidence-based treatments. Within families, socioecological stress may impact developmental trajectories from pregnancy through adulthood. Caregivers' wellbeing and stress levels, parenting practices, and competence in promoting positive identity may influence youths' development of accurate appraisal strategies and positive coping skills to protect them from stress. Families with effective communication strategies to discuss community strengths, navigate through stressful encounters, and build self-esteem may be more likely to buffer the effects of stress on their children's development. Although evidence-based trauma treatments to address the effects of child abuse and neglect, such as Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), have demonstrated efficacy in reducing symptoms of posttraumatic stress (PTSD) broadly speaking, they are not designed to address the specific challenges that youth from socioecological contexts with multiple risk factors along with child abuse and neglect experiences face in counteracting both PTSD and additional stress. Novel approaches are being developed that can support families in building socialization skills. This pilot study examines the feasibility and acceptability of augmenting TF-CBT with socialization practices to improve outcomes for youth ages 10-15 who have experienced child abuse and neglect and their families by supporting parenting strategies. A RE-AIM/PRISM framework (including Reach, Effectiveness, Adoption, Implementation, and Maintenance with emphasis on contextual factors at multiple levels of the implementation setting) is incorporating stakeholder perspectives and evaluating the enhanced version of TF-CBT compared with current practices, while identifying barriers and facilitators to implementation to guide future larger-scale trials. Developing interventions to support parenting strategies that can promote positive socialization and identity for youth facing the combined effects of child abuse and neglect and socioecological stress is of high public health significance. Given the lifelong cascades that accompany child abuse and neglect and discrimination, determining best practices for improving behavioral health outcomes for youth who have experienced child abuse and neglect is highly significant.

This Resilient Roots Pilot is integrated into the TRANSFORM Center on Child Abuse and Neglect to promote translation of research findings into clinical interventions, to inform the next generation of research on child abuse and neglect, and to facilitate dissemination of research and practice knowledge/skills to varied stakeholders. The research utilizes a developmental psychopathology perspective, incorporating multiple methods within a lifespan framework and implementation science approach. Exposure to child abuse and neglect frequently results in long-term detrimental effects on mental health. Interventions to address specific socioecological stress for symptomatic youth receiving human centered mental health services are lacking, and use of mental health services that are acceptable to families are too often misaligned with their representation in the population in general and overrepresentation in the child welfare system specifically. Incorporating support for families in enhancing socialization and coping skills specific to addressing contextual stress and trauma has relevance for public health. Although TF-CBT is an evidence-based treatment for children who have experienced trauma, determining best practices for implementing enhanced TF-CBT with socialization components is urgently needed to address these gaps and provide optimal intervention.

The study Aims for the full project are as follows:

Aim 1: From a community-based participatory research framework, engage community partners and assess acceptability of augmenting TF-CBT for youth ages 10-15, as well as to inform study design, and implementation via focus groups with diverse stakeholders (youth, family, mental health clinicians) to inform Aim 2.

Aim 2: Evaluate the feasibility of a pilot randomized control trial testing the augmentation of TF-CBT to improve coping and socialization, and to reduce mental health symptoms in youth with CAN histories.

Aim 3: Investigate whether TF-CBT leads to greater improvement in mental health symptoms for youth with CAN when augmented with addressing socioecological stresses.

ELIGIBILITY:
Inclusion Criteria:

Youth participants will be:

* Youth who are seeking services at the University of Rochester Medical Center Pediatric Behavioral Health and Wellness and whose caregivers consent to participate and youth assent to participate.
* Youth ages 10-15 years at the time of enrollment.
* Youth with histories of child maltreatment as determined by screening positive on at least 1 child abuse or neglect item from the ACE scale completed by caregiver report and/or report of child trauma exposure during the phone screen at intake or on the Child PTSD Symptom Checklist assessment tool completed independently by youth.

Exclusion Criteria:

* Significant cognitive limitations or psychiatric condition that would interfere with ability to participate in the assessment and treatment portions of the study
* Physical disability, if we do not have a way of providing necessary accommodations to allow them to engage in the study
* Youth in foster care or residential treatment
* Caregivers with self-reported significant psychiatric needs or substance use requiring inpatient treatment that would interfere with their ability to participate in the assessment and treatment of study
* Language: English speaking proficiency that precludes completing assessment measures

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Symptoms | Assessed at pre- and post-intervention (following 12-25 sessions), approximately 6 months later
  Change in symptoms of posttraumatic stress as measured by Child Posttraumatic Stress Disorder Symptom Checklist (Child Report). Lower scores indicate lower symptoms of posttraumatic stress (range 0-80).

SECONDARY OUTCOMES:
Patient Perceptions of Treatment | Assessed at intervention completion (following 12-25 sessions), approximately 6 months after enrollment
  Participant satisfaction with intervention assessed through a Client Satisfaction Questionnaire, 4 point scale that will be scored with reverse scoring on some items such that higher scores are reflective of higher satisfaction, range 9-36
Provider Perceptions of Treatment | Assessed at intervention completion (following 12-25 sessions), approximately 6 months after enrollment
  Clinician satisfaction with intervention assessed through Clinician Evaluation Questionnaire, with 7-point scale with higher scores indicating more agreement across domains of knowledge, confidence, intentions, consequences, resources, social influences, priorities, intervention characteristics, and memory
Participant attendance and participation in treatment | Assessed at intervention completion (following 12-25 sessions), approximately 6 months after enrollment
  Number of sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
The study will share de-identified data using NICHD Data Specimen Hub (DASH).